CLINICAL TRIAL: NCT01840059
Title: A Randomised Controlled Trial Investigating the Effect of Transcatheter Renal Sympathetic Denervation on Symptoms and Cardiac Function in Patients With Heart Failure With Preserved Ejection Fraction.
Brief Title: Renal Denervation in Heart Failure With Preserved Ejection Fraction
Acronym: RDT-PEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012HS001B
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Cardiac Failure
Keywords: Cardiac Failure; Autonomic Denervation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal sympathetic denervation (Experimental): Renal denervation using the Medtronic Symplicity catheter.
  Interventions: Device: Renal sympathetic denervation
- Control (No Intervention): HF-PEF patients who will serve as control.

INTERVENTIONS:
Device: Renal sympathetic denervation — A fit for purpose radiofrequency catheter is guided to the renal artery using fluoroscopy. This is connected to an external RF generator. RF energy is applied through the catheter to the renal artery wall with the goal of disrupting the sympathetic nerves which run in the adventitia
  Other Names: Medtronic Symplicity Catheter
  Arms: Renal sympathetic denervation

SUMMARY:
The purpose of this study is to determine whether renal sympathetic denervation (RSD)(a treatment that lowers the activity of the sympathetic nervous system) is useful in the management of patients with heart failure with preserved ejection fraction (HF-PEF).

DETAILED DESCRIPTION:
Increasing evidence suggests an important role of activation of the sympathetic nervous system (SNS) in heart failure with preserved left ventricular ejection fraction. The current study aims to evaluate efficacy of renal sympathetic denervation for the modulation of the SNS in patients with HF-PEF.

ELIGIBILITY:
Inclusion Criteria:

* EF>40%
* NHYA 2-3
* Evidence of HF-PEF (mixture of dilated left atrium, left ventricular hypertrophy, raised E/E', elevated LVEDP/PCWP, raised BNP)

Exclusion Criteria:

* Previously documented EF<40%
* Hypertrophic, restrictive, dilated cardiomyopathy
* Significant valvular heart disease
* Unfavourable renal artery anatomy for renal denervation
* eGFR<45
* Contraindication to MRI
* Myocardial infarction, unstable angina or cerebrovascular accident in last 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Symptoms | 12 months
  Minnesota Living with Heart Failure Questionnaire
Change in Exercise Function | 12 months
  Peak VO2 (Oxygen Uptake) on cardiopulmonary exercise testing
Change in Heart Failure Biomarker | 12 months
  BNP (Natriuretic peptide)
Change in LV (Left Ventricle) filling pressure | 12 months
  E/E' on echocardiography
Change in LV remodelling | 12 months
  LV mass index
Change in Left atrial (LA) size | 12 months
  LA volume index

SECONDARY OUTCOMES:
Change in Autonomic function | 3 and 12 months
  Heart rate variability
Change in Renal function | 3 and 12 months
  Urea and Creatinine
Change in Vascular function | 3 and 12 months
  Aorta MRI (Magnetic Resonance Imaging)
Change in Autonomic function | 3 and 12 months
  mIBG radiotracer assessment
Change in neurohormones | 3 and 12 months
  Neurohormones
Change in renal blood flow | 3 and 12 months
  Renal MRI
Change in Blood pressure | 3 and 12 months
  ABPM (Ambulatory Blood Pressure Monitoring)
Change in Endothelial function | 3 and 12 months
  EndoPat

CONTACTS AND LOCATIONS:
Overall Officials: Carlo di Mario, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Background] Sobotka PA, Krum H, Bohm M, Francis DP, Schlaich MP. The role of renal denervation in the treatment of heart failure. Curr Cardiol Rep. 2012 Jun;14(3):285-92. doi: 10.1007/s11886-012-0258-x. PMID 22392370